CLINICAL TRIAL: NCT06416670
Title: Skilled Nursing Facility Care at Home: A Randomized Controlled Trial
Brief Title: Skilled Nursing Facility Care at Home
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston Medical Center (Other); Cambridge Health Alliance (Other)
Responsible Party: Principal Investigator, David Levine, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024P000266
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Skilled Nursing Facility; Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual skilled nursing facility care (No Intervention): Control subjects will receive care at a skilled nursing facility as per usual.
- Rehab at home (Active Comparator): Intervention subjects will receive care in their home from a specialized care team.
  Interventions: Other: Skilled nursing facility care at home

INTERVENTIONS:
Other: Skilled nursing facility care at home — Skilled nursing facility care at home delivers a range of advanced rehabilitation services in patients' homes, enabling care at home despite requiring intensive rehabilitative care. Our approach blends personalized, high-level professional care with innovative technology applications to ensure adequate rehabilitation.
  Arms: Rehab at home

SUMMARY:
We will perform a parallel-group multicenter patient-level randomized controlled evaluation of skilled nursing facility care at home. Patients typically referred to a skilled nursing facility following hospitalization will be eligible for enrollment. Instead of admission to a skilled nursing facility, participants will receive care from a technology-enabled team in their own homes or will be allocated to receive care in a traditional skilled nursing facility setting.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years old
* Requires SNF PAC care following hospitalization, as determined by the inpatient team (requires documented rehabilitative therapy recommendation)
* Community-dwelling before hospitalization
* Likely to return to community-dwelling status following short-term rehabilitation as determined by RAH liaison
* Lives within 10 miles of any study site hospital (or per specified catchment)
* Surgical trauma and elective patients (weight bearing as tolerated and transfer with no more than one-person assist)
* Neurology patients - Stroke (needs acute rehabilitation, but insurance will not cover, so bound for SNF. Does not meet acute rehabilitation criteria and does not need long-term placement)

Exclusion Criteria:

* Environmental

  * Undomiciled
  * No working heat (October-April), no working air conditioning if forecast > 80°F, or no running water
  * In police custody
  * Resides in a facility that does not allow advanced on-site care
  * Domestic violence screen positive
  * Weapons that cannot be appropriately secured
  * Difficulty accessing the bathroom (unless there is space for a bedside commode where the patient sleeps or if the patient is entirely dependent on toileting)
  * Home has insufficient accessible space to sleep, eat, and perform rehabilitative therapy
  * Home lacks sufficient kitchen facilities to either cook or heat meals
  * Patient, or patient's family caregiver, unable to communicate via telephone
  * Patient, or patient's family caregiver, lacks consistent access to a telephone
* Clinical

  * Requires more than one assist (unless the family can provide additional 24/7 assistance)
  * Requires care of new ostomy or teaching ostomy care
  * Requires frequent suctioning, tracheostomy, and ventilator needs
  * Requires total parenteral nutrition
  * Requires nasogastric tube feeds
  * Requires durable medical equipment not already in place at home and excluded below
  * Requires daily subcutaneous injection unless patient or family caregiver is teachable and able to administer daily
  * Acute delirium noted by RAH liaison requiring more than one caregiver
  * Active psychiatric diagnosis without an adequate treatment plan
  * On methadone requiring daily pickup of medication
  * Requires administration of intravenous controlled substances
  * Requires administration of specialty medications not already in place at home
  * Requires transfusion of blood products
  * Requires three times weekly or more transfers back and forth to obtain specialty medical care
  * Requires hemodialysis
  * Orthopedic trauma and elective patients
  * Traumatic brain injury
  * Wound or appliance care that requires daily nursing care
  * For spine trauma: neurologic deficits requiring more than one assist
* Neurology patients

  * PRESS score (for ischemic stroke; use PRESS app): no return to pre-stroke diet > 50%
  * FUNC score (for primary intracerebral hemorrhage only): <75% probability of functional independence at 90 days
  * ASTRAL score (for ischemic stroke only and patients with pre-stroke independence [Modified Rankin Scale 0-2]): <75% probability of a 90-day poor functional outcome (Modified Rankin Scale result of 3-6)
* RAH census is full

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in activities of daily living between admission to rehab and discharge from rehab | Admission to rehab until discharge from rehab, no more than 6 months
  Subtract the patient's activities of daily living at discharge from rehab from the patient's activities of daily living on admission to rehab.

SECONDARY OUTCOMES:
Percent time supine per day | Admission to rehab until discharge from rehab, no more than 6 months
  The percentage of time a patient is supine per day, as measured by their wrist-worn accelerometer.
Total direct medical expenditure | Admission to rehab until discharge from rehab, no more than 6 months
  The percent difference in direct cost of care to deliver rehab care.
Patient experience with care | Admission to rehab until discharge from rehab, no more than 6 months
  The Picker patient experience questionaire-15
30-day readmission or 30-day mortality | Discharge from rehab until 30-days later, no more than 30-days
  The percentage of patients who are readmitted or deceased within 30-days of discharge from rehab.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts
  - Cambridge Health Alliance, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: No